CLINICAL TRIAL: NCT01745718
Title: Targeted Biopsies and the Role of Cytological Imprints for Diagnosis of Prostate Cancer
Brief Title: Clinical Study Evaluating Targeted Biopsies and Cytological Imprints in Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped for technical reasons
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OsloUH_2
Record Dates: First submitted 2012-11-20; First posted 2012-12-10 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; targeted biopsies; cytological imprints; histology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI and targeted biopsies (Other): All patients receive the same level/number of diagnostic procedures. They all undergo targeted biopsies which are compared to the cytological imprints.
  Interventions: Other: Cytological imprints

INTERVENTIONS:
Other: Cytological imprints — Each targeted biopsy is subject to cytological imprints. It causes no extra biopsies or extra discomfort for the patients

SUMMARY:
The investigators will evaluate the accuracy of performing cytological imprints of targeted biopsies when diagnosing prostate cancer.

It is useful to know whether the biopsy is cancer or not, in order to know when to stop sampling and when to continue.

The strategy is used in other types of cancer, e.g lung, breast etc

DETAILED DESCRIPTION:
Background:

When substituting a random biopsy procedure with a few targeted biopsies, it is of outmost importance to know immediately if the biopsy is positive or not. A recent study has demonstrated a high sensitivity and specificity of imprint cytology of random biopsies.

Aim:

The correlation between cytological imprints and histology of targeted prostate biopsies

Material&Method:

All patients in this study are already participating in an ongoing randomized biopsy study (NCT01455792) comparing:

1. Preoperative MRI and targeted biopsies + random biopsies .
2. Random biopsies (gold standard).

Only patients with a positive MRI were included in this collateral study.

The cytological imprints (negative/positive) of each targeted biopsy is compared to the histology (negative/positive) and Gleason score.

ELIGIBILITY:
Inclusion Criteria:

* Prostate specific antigene (PSA) 4-20ng/ml, and/or abnormal digital rectal examination
* No previous prostate biopsies
* Positive MRI
* Signed letter of informed concent

Exclusion Criteria:

* Contraindications to MRI
* Previous prostate biopsies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The rate of positive and negative cytological imprints, e.g presence of malignant cells or not. | 15 months
  The cytological imprints will be compared to the histology of targeted biopsies (defined as gold standard). Measure of agreement, sensitivity and specificity will be calculated.

SECONDARY OUTCOMES:
Interobserver variability | 15 months
  The cytological imprints will be evaluated by three different cytologists and classified as either negative or positive. The results will be compared to the histology which defines the gold standard. Any difference in evaluation will be assessed.

OTHER OUTCOMES:
The detection rate of high grade cancer | 15 months
  The cytology will be compared to the specific Gleason score in patients with positive histology in order to evaluate any difference in the detection rate of intermediate/high grade cancer (Gleason score 7 or higher) and low grade cancer (<Gleason score 6).

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Baco, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital , Aker, Oslo, Norway